CLINICAL TRIAL: NCT00704847
Title: A Randomized, Double-Blind, Multi-Center, Placebo-Controlled Study to Evaluate the Efficacy and Safety of Oral Salmon Calcitonin in the Treatment of Subjects With Knee Osteoarthritis
Brief Title: Efficacy and Safety of Oral Salmon Calcitonin in Patients With Knee Osteoarthritis (OA 2 Study)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Male subjects were terminated due to an imbalance in prostate cancer events
Sponsor: Nordic Bioscience A/S (Industry)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CSMC021C2302
Record Dates: First submitted 2008-06-24; First posted 2008-06-25 (Estimated); Results first posted 2012-09-12 (Estimated); Last update posted 2019-04-24 (Actual); Status verified 2019-04

CONDITIONS: Osteoarthritis
Keywords: Osteoarthritis, oral salmon calcitonin, treatment, efficacy,; tolerability
MeSH Terms: conditions — Osteoarthritis | interventions — salmon calcitonin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): SMC021 Oral Calcitonin
  Interventions: Drug: Oral Salmon Calcitonin
- 2 (Placebo Comparator): SMC021 Placebo
  Interventions: Drug: Oral Salmon Calcitonin (Placebo)

INTERVENTIONS:
Drug: Oral Salmon Calcitonin — 0.8mg SMC021, twice daily
  Arms: 1
Drug: Oral Salmon Calcitonin (Placebo) — 0.8mg Placebo, twice daily
  Arms: 2

SUMMARY:
The purpose of this phase III study is to Evaluate the Efficacy and Safety of Oral Salmon Calcitonin in the Treatment of Patients with Osteoarthritis of the Knee

ELIGIBILITY:
Inclusion Criteria:

* Medical history and symptoms of knee osteoarthritis

Exclusion Criteria:

* Any other disease or medication affecting the bone or cartilage.
* Any clinical signs or laboratory evidence diseases, which in the Investigator's opinion would preclude the participant from adhering to the Protocol or completing the trial.

Other protocol defined inclusion/exclusion criteria may apply

Ages: 51 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1030 (Actual)
Dates: Start 2008-06; Primary Completion 2011-05 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bente Juel Riis, MD, Study Director — Nordic Bioscience
Locations (18):
- United States (6):
  - Achieve Clinical Research, LLC, Tuscaloosa, Alabama
  - Center for Healthy Aging, Sacramento, California
  - Northwestern Center for Clinical Research, Chicago, Illinois
  - Midwest Pharmaceutical Research, City of Saint Peters, Missouri
  - Thurston Arthritis Research Center, Chapel Hill, North Carolina
  - Rheumatology Clinical Research Unit, Beachwood, Ohio
- Hospital Universitaire St. Luc, UCL 5390, Brussels, Belgium
- Centre de Rhumatologie St-Louis, Sainte-Foy (Québec), Canada
- CCBR Czech, Pardubice, Czechia
- Denmark (3):
  - CCBR Aalborg, Aalborg
  - CCBR Ballerup, Ballerup Municipality
  - CCBR Vejle, Vejle
- CCBR Hong Kong, Hong Kong, Hong Kong
- Poland (2):
  - Centrum Osteoporozy i Chorób Kostno Stawowych, ul. Waryńskiego 6/2, Bialystok
  - CCBR Poland, Warsaw
- CCBR Romania, Bucharest, Romania
- Hospital Universitario de la Paz, Madrid, Spain
- Little Common Surgery, Bexhill-on-Sea, East Sussex, United Kingdom

REFERENCES:
- [Derived] Bihlet AR, Bjerre-Bastos JJ, Andersen JR, Byrjalsen I, Karsdal MA, Bay-Jensen AC. Clinical and biochemical factors associated with risk of total joint replacement and radiographic progression in osteoarthritis: Data from two phase III clinical trials. Semin Arthritis Rheum. 2020 Dec;50(6):1374-1381. doi: 10.1016/j.semarthrit.2020.03.002. Epub 2020 Mar 15. PMID 32249039
- [Derived] Bihlet AR, Byrjalsen I, Bay-Jensen AC, Andersen JR, Christiansen C, Riis BJ, Karsdal MA. Associations between biomarkers of bone and cartilage turnover, gender, pain categories and radiographic severity in knee osteoarthritis. Arthritis Res Ther. 2019 Sep 3;21(1):203. doi: 10.1186/s13075-019-1987-7. PMID 31481084
- [Derived] Bihlet AR, Byrjalsen I, Bay-Jensen AC, Andersen JR, Christiansen C, Riis BJ, Valter I, Karsdal MA, Hochberg MC. Identification of pain categories associated with change in pain in patients receiving placebo: data from two phase 3 randomized clinical trials in symptomatic knee osteoarthritis. BMC Musculoskelet Disord. 2018 Jan 17;19(1):17. doi: 10.1186/s12891-018-1938-5. PMID 29343266
- [Derived] Karsdal MA, Byrjalsen I, Alexandersen P, Bihlet A, Andersen JR, Riis BJ, Bay-Jensen AC, Christiansen C; CSMC021C2301/2 investigators. Treatment of symptomatic knee osteoarthritis with oral salmon calcitonin: results from two phase 3 trials. Osteoarthritis Cartilage. 2015 Apr;23(4):532-43. doi: 10.1016/j.joca.2014.12.019. Epub 2015 Jan 9. PMID 25582279
- [Derived] Henriksen K, Bay-Jensen AC, Christiansen C, Karsdal MA. Oral salmon calcitonin--pharmacology in osteoporosis. Expert Opin Biol Ther. 2010 Nov;10(11):1617-29. doi: 10.1517/14712598.2010.526104. Epub 2010 Oct 11. PMID 20932224

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were enrolled at 18 centers in 10 countries: 6 centers in the US, 1 center in the UK, 1 center in Spain,1 center in the Czech Republic, 3 centers in Denmark, 1 center in Hong Kong, 2 centers in Poland, 1 center in Romania, 1 center in Belgium and 1 center in Canada.
  First patient randomized: 1 Aug 08 Last patient visit: 10 May 2011
Groups:
- SMC021 Oral Calcitonin: 0.8 mg SMC021 Oral Calcitonin twice daily
- SMC021 Placebo: 1 SMC021 Placebo tablet twice daily
Period: Overall Study
Arm/Group | SMC021 Oral Calcitonin | SMC021 Placebo
Started | 521 | 509
Completed | 300 | 339
Not Completed | 221 | 170

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SMC021 Oral Calcitonin | SMC021 Placebo | Total
Number analyzed (Participants) | 521 | 509 | 1030
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 292 | 288 | 580
  >=65 years | 229 | 221 | 450
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.4 (7.0) | 64.2 (6.8) | 64.3 (6.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 321 | 305 | 626
  Male | 200 | 204 | 404
Region of Enrollment [Number; unit: participants]
  United States | 26 | 21 | 47
  Hong Kong | 72 | 72 | 144
  Czech Republic | 36 | 35 | 71
  Canada | 11 | 8 | 19
  Spain | 4 | 2 | 6
  Belgium | 7 | 7 | 14
  Poland | 67 | 66 | 133
  Romania | 9 | 9 | 18
  Denmark | 263 | 264 | 527
  United Kingdom | 26 | 25 | 51

OUTCOME MEASURES:

1. Primary Outcome: Joint Space Width (JSW) in the Medial Tibia-femoral Knee Joint in the Signal Knee Measured by X-ray Change From Baseline Over 24 Months
Description: The signal knee was chosen prior to randomization based on which knee met the inclusion and exclusion criteria. The JSW is the space measured in mm between the 2 bones in the knee joint and this is assessed by x-ray. The JSW decreases with disease progression. The lower limit for participation in the trial were 2 mm JSW. There were no upper limit as long as inclusion and exclusion criteria were met. The outcome was measured as a change in JSW from baseline to month 24.
Time Frame: Change from baseline to 24 months
Population: The number of participants analysed for this outcome is the intent-to-treat (ITT) population. ITT is the number of randomized subjects who received at least one dose of study medication. There were 2 patients in the randomized population who did not receive any study drug and where therefore excluded from the ITT analysis.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | SMC021 Oral Calcitonin | SMC021 Placebo
Number analyzed (Participants) | 520 | 508
mm | -0.32 (0.693) | -0.40 (0.768)

2. Primary Outcome: Pain Subscore Change From Baseline Over 24 Months as Assessed by Western Ontario and McMaster Universities Arthritis (WOMAC) Index
Description: WOMAC is a self-administered set of standardized questionnaires to evaluate the condition of patients with osteoarthritis of the knee. The subject marks on a scale (1-100) the pain associated with performing each daily activity listed in the questionnaire. 0 is no pain (best), 100 is extreme pain (Worst). The total pain sub score for the questions are then calculated. Total possible minimum sub score is 0, maximum is 500. The final outcome is the absolute change from baseline to 24 months. If the outcome is less that 0 there is improvement (less pain).
Time Frame: Change from baseline to 24 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | SMC021 Oral Calcitonin | SMC021 Placebo
Number analyzed (Participants) | 520 | 508
Units on a scale | -80.6 (112.22) | -87.9 (116.25)

3. Secondary Outcome: Bone & Cartilage Metabolism Biochemical Marker Change (Percentage).
Description: The central laboratory analyzed serum CTX-I (S-Crosslaps, Elecsys) and osteocalcin as well as urine CTX I/creatinine and CTX-II/creatinine. These biomarkers were analysed in order to assess the cartilage and bone turonver ratio to baseline at month 24.
Time Frame: From baseline to 24 months
Population: The number of participants analysed for these outcomes were a total of 150 subjects from the intent-to-treat (ITT) population evenly distributed across sites, all with completed baseline as well as all follow-up visits.
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | SMC021 Oral Calcitonin | SMC021 Placebo
Number analyzed (Participants) | 69 | 81
percentage of change
  Serum CTX-I (ng/mL): number analyzed (Participants) | 68 | 81
  Serum CTX-I (ng/mL) | 50.6 (83.74) | 40.6 (45.52)
  Serum Osteocalcin (ng/mL): number analyzed (Participants) | 68 | 81
  Serum Osteocalcin (ng/mL) | 3.6 (37.42) | 3.9 (26.32)
  24-h urine CTX-I/creatinine (µg/mmol): number analyzed (Participants) | 69 | 79
  24-h urine CTX-I/creatinine (µg/mmol) | 9.8 (85.95) | 7.2 (44.36)
  24-h urine CTX-II/creatinine (ng/mmol): number analyzed (Participants) | 69 | 79
  24-h urine CTX-II/creatinine (ng/mmol) | 2.6 (63.13) | 2.3 (51.07)

4. Secondary Outcome: Knee Disease Progression Assessed by MRI
Description: Knee cartilage volume and thickness was assessed by MRI in patients from the sites in Ballerup, Denmark, the Czech Republic, and Romania using a quality controlled low-field 0.18T C-Span scanner from Esaote dedicated to the imaging of extremities. The same solenoid coil was used for all patients at a given site.
Time Frame: From baseline to month 12 and month 24
Population: Subset of patients from the sites in Ballerup (Denmark), Czech Republic and Romania
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | SMC021 Oral Calcitonin | SMC021 Placebo
Number analyzed (Participants) | 152 | 149
percentage of change
  Cartilage Volume Month 12: number analyzed (Participants) | 115 | 130
  Cartilage Volume Month 12 | 3.4 (9.11) | 3.0 (13.16)
  Cartilage Volume Month 24: number analyzed (Participants) | 103 | 119
  Cartilage Volume Month 24 | 2.6 (10.18) | 3.5 (12.73)
  Cartilage Thickness Month 12: number analyzed (Participants) | 115 | 130
  Cartilage Thickness Month 12 | 4.7 (10.64) | 4.7 (8.24)
  Cartilage Thickness Month 24: number analyzed (Participants) | 103 | 119
  Cartilage Thickness Month 24 | 4.5 (10.78) | 4.1 (8.67)

5. Secondary Outcome: Questionnaire to Assess Function and Physical Activity
Description: Function and physical activity were assessed by assessed by WOMAC function sub-score in the signal knee. The criteria for assessment of the functional classification according to the American Rheumatism Association (ARA) were as follows (Hochberg et al 1992):
  I. Completely able to perform usual activities of daily living (self-care, vocational and avocational) II. Able to perform usual self-care and vocational activities, but limited in avocational activities.
  III. Able to perform usual self-care activities, but limited in vocational and avocational activities.
  IV. Limited ability to perform usual self-care activities, vocational and avocational activities.
  Self-care activities included dressing, feeding, bathing, grooming, and toileting. Avocational (recreational and/or leisure) and vocational (work, school, homemaking) activities were patient-desired and age- and sex-specific.
Time Frame: From baseline to months 1, 6, 12 and 24
Population: The number of participants analysed for this outcome is the intent-to-treat (ITT) population. ITT is the number of randomized subjects who received at least one dose of study medication.
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | SMC021 Oral Calcitonin | SMC021 Placebo
Number analyzed (Participants) | 520 | 508
percentage of change
  Month 1: number analyzed (Participants) | 489 | 495
  Month 1 | -4.8 (44.89) | -1.9 (131.20)
  Month 6: number analyzed (Participants) | 437 | 452
  Month 6 | -22.6 (49.03) | -17.9 (64.15)
  Month 12: number analyzed (Participants) | 386 | 416
  Month 12 | -28.0 (53.97) | -28.4 (59.79)
  Month 24: number analyzed (Participants) | 336 | 370
  Month 24 | -30.3 (77.51) | -25.1 (143.05)

6. Secondary Outcome: Questionnaire to Assess Stiffness in the Signal Knee.
Description: WOMAC's stiffness subscore was used to assess the stiffness in the signal knee. WOMAC is a self-administered set of standardized questionnaires to evaluate the condition of patients with osteoarthritis of the knee. The subject marks on a scale (1-100) the degree of joint stiffness for when performing each daily function listed in the questionnaire. 0 is no stiffness (best), 100 is extreme stiffness (worst). The total function sub score for the questions are then calculated. Total possible minimum sub score is 0, maximum is 200. The final outcome is the absolute change from baseline to 24 months. If the outcome is less that 0 there is improvement (less stiffness).
  Patients were instructed not to take analgesics for 3 days prior to the WOMAC test.
Time Frame: Baseline to month 24
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | SMC021 Oral Calcitonin | SMC021 Placebo
Number analyzed (Participants) | 520 | 508
percentage of change | -26.1 (90.88) | -20.3 (179.22)

7. Secondary Outcome: Questionnaire to Assess Health-related Quality of Life
Description: Health-related quality of life was assessed by the EQ-5D questionnaire, which is a patient questionnaire for measure of health, developed by the EuroQol Group.The EQ-5D questionnaire was administered to patients in order to measure change in health-related quality of life (HRQoL) over 2 years.
  The subjects marks on a VAS scale from 0 to 100 the number that best describes their health today (0 is worst imaginable health state and 100 is best imaginable health state).
  The change from baseline in the EQ-5D VAS was calculated.
Time Frame: From baseline to month 24
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | SMC021 Oral Calcitonin | SMC021 Placebo
Number analyzed (Participants) | 515 | 504
percentage of change | 13.70 (38.763) | 11.82 (40.645)

8. Secondary Outcome: Questionnaire to Assess Pain
Description: Pain was assessed by the WOMAC subscore in the signal knee by visit. Patients assessed their current pain level using a 100 mm visual analogue scales (VAS) by placing an X on the line that best describes his/her pain, where 0 equaled "No Pain" and 100 equaled "Worst Pain Imaginable". Patients were instructed not to take analgesics for 3 days prior to the VAS.
Time Frame: Baseline, month 1, month 6, month 12, month 24
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | SMC021 Oral Calcitonin | SMC021 Placebo
Number analyzed (Participants) | 520 | 508
percentage of change
  Month 1: number analyzed (Participants) | 489 | 495
  Month 1 | -6.7 (49.50) | -9.1 (45.26)
  Month 6: number analyzed (Participants) | 438 | 452
  Month 6 | -26.9 (51.73) | -26.9 (50.43)
  Month 12: number analyzed (Participants) | 386 | 416
  Month 12 | -31.0 (68.05) | -34.6 (61.30)
  Month 24: number analyzed (Participants) | 336 | 370
  Month 24 | -35.1 (91.63) | -37.1 (77.55)

ADVERSE EVENTS:
Time Frame: From baseline to 30 days following the end of participation
Description: The safety population is all patients randomized who received at least one dose of study medication. There were 2 patients in the randomized population who did not receive any study drug and where therefore excluded from the safety analysis.
Arm/Group | SMC021 Oral Calcitonin | SMC021 Placebo
Serious Adverse Events (participants affected / at risk) | 77/520 | 80/508
Other Adverse Events (participants affected / at risk) | 474/520 | 459/508
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SMC021 Oral Calcitonin (N=520) | SMC021 Placebo (N=508)
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Splenomegaly (Blood and lymphatic system disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 2 | 3
Angina pectoris (Cardiac disorders) | 3 | 0
Acute myocardial infarction (Cardiac disorders) | 2 | 0
Myocardial infarction (Cardiac disorders) | 0 | 2
Myocardial ischaemia (Cardiac disorders) | 1 | 1
Acute coronary syndrome (Cardiac disorders) | 1 | 0
Arrhythmia (Cardiac disorders) | 0 | 1
Atrioventricular block (Cardiac disorders) | 0 | 1
Cardiac arrest (Cardiac disorders) | 1 | 0
Coronary artery disease (Cardiac disorders) | 0 | 1
Coronary artery thrombosis (Cardiac disorders) | 0 | 1
Sinus arrhythmia (Cardiac disorders) | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 1 | 0
Middle ear inflammation (Ear and labyrinth disorders) | 1 | 0
Goitre (Endocrine disorders) | 1 | 1
Hyperparathyrodism (Endocrine disorders) | 0 | 1
Optic ischaemic neuropathy (Eye disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 1
Gastritis (Gastrointestinal disorders) | 2 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 2
Abdominal hernia (Gastrointestinal disorders) | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Crohn´s disease (Gastrointestinal disorders) | 0 | 1
Diverticulum intestinal (Gastrointestinal disorders) | 0 | 1
Gastrointestinal inflammation (Gastrointestinal disorders) | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Chest pain (General disorders) | 1 | 1
Foreign body reaction (General disorders) | 1 | 0
Pyrexia (General disorders) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 2 | 1
Cholangitis acute (Hepatobiliary disorders) | 1 | 1
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Jaundice (Hepatobiliary disorders) | 1 | 0
Hypersensitivity (Immune system disorders) | 0 | 2
Bronchitis (Infections and infestations) | 0 | 2
Cellulitis (Infections and infestations) | 1 | 1
Pneumonia (Infections and infestations) | 0 | 2
Urinary tract infection (Infections and infestations) | 1 | 1
Diverticulitis (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 1
Infection (Infections and infestations) | 1 | 0
Orchitis (Infections and infestations) | 0 | 1
Pancreatic abscess (Infections and infestations) | 0 | 1
Sinusitis (Infections and infestations) | 0 | 1
Wrist fracture (Injury, poisoning and procedural complications) | 1 | 2
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 1
Femur fracture (Injury, poisoning and procedural complications) | 2 | 0
Radius fracture (Injury, poisoning and procedural complications) | 0 | 2
Tibia fracture (Injury, poisoning and procedural complications) | 1 | 1
Abdominal injury (Injury, poisoning and procedural complications) | 0 | 1
Chemical peritonitis (Injury, poisoning and procedural complications) | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 1
Cystitis radiation (Injury, poisoning and procedural complications) | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 1 | 0
Ligament rupture (Injury, poisoning and procedural complications) | 0 | 1
Multiple fractures (Injury, poisoning and procedural complications) | 1 | 0
Open wound (Injury, poisoning and procedural complications) | 1 | 0
Overdose (Injury, poisoning and procedural complications) | 1 | 0
Patella fracture (Injury, poisoning and procedural complications) | 0 | 1
Postoperative hernia (Injury, poisoning and procedural complications) | 0 | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 1
Prostatic specific antigen increased (Investigations) | 2 | 3
Hypernatraemia (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 | 6
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 4 | 8
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 3 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 1
Arthritis reactive (Musculoskeletal and connective tissue disorders) | 1 | 0
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Foot deformity (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 5
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0
Abdominal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Morton´s neuroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Multiple myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Prostatic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 2 | 0
Amytrophic lateral sclerosis (Nervous system disorders) | 1 | 0
Cauda equina syndrome (Nervous system disorders) | 0 | 1
Cerebral thrombosis (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0
Sciatica (Nervous system disorders) | 1 | 0
Spondylitic myelopathy (Nervous system disorders) | 1 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 1 | 0
Trigeminal neuralgia (Nervous system disorders) | 0 | 1
Alcohol withdrawal syndrome (Psychiatric disorders) | 1 | 0
Depression (Psychiatric disorders) | 1 | 0
Stress urinary incontinence (Renal and urinary disorders) | 1 | 1
Urethral stenosis (Renal and urinary disorders) | 0 | 1
Urinary bladder polyp (Renal and urinary disorders) | 1 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 | 1
Prostatitis (Reproductive system and breast disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Diaphragmatic hernia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1
Joint prosthesis user (Social circumstances) | 0 | 1
Hip arthroplasty (Surgical and medical procedures) | 1 | 1
Knee arthroplasty (Surgical and medical procedures) | 1 | 1
Aortic surgery (Surgical and medical procedures) | 1 | 0
Cataract operation (Surgical and medical procedures) | 1 | 0
Joint arthroplasty (Surgical and medical procedures) | 1 | 0
Joint stabilisation (Surgical and medical procedures) | 0 | 1
Circulatory collapse (Vascular disorders) | 1 | 0
Thrombosis (Vascular disorders) | 0 | 1
Venous stenosis (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | SMC021 Oral Calcitonin (N=520) | SMC021 Placebo (N=508)
Arthralgia (Musculoskeletal and connective tissue disorders) | 86 | 111
Hot flush (Vascular disorders) | 88 | 22
Back Pain (Musculoskeletal and connective tissue disorders) | 52 | 54
Nausea (Gastrointestinal disorders) | 77 | 15
Influenza (Infections and infestations) | 46 | 40
Nasopharyngitis (Infections and infestations) | 34 | 39
Diarrhoea (Gastrointestinal disorders) | 45 | 27
Hypertension (Vascular disorders) | 31 | 39
Dyspepsia (Gastrointestinal disorders) | 48 | 21
Headache (Nervous system disorders) | 26 | 27
Pain in extremity (Musculoskeletal and connective tissue disorders) | 27 | 23
Dizziness (Nervous system disorders) | 32 | 17
Hypercholesterolaemia (Metabolism and nutrition disorders) | 24 | 24
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 26 | 20
Upper respiratory tract infection (Infections and infestations) | 20 | 23
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 14 | 25
Pneumonia (Infections and infestations) | 20 | 15
Abdominal pain upper (Gastrointestinal disorders) | 19 | 15
Cystitis (Infections and infestations) | 13 | 21
Viral infection (Infections and infestations) | 16 | 18
Cough (Respiratory, thoracic and mediastinal disorders) | 16 | 15
Oedema peripheral (General disorders) | 17 | 14
Bronchitis (Infections and infestations) | 19 | 11
Procedural pain (Injury, poisoning and procedural complications) | 10 | 20
Influenza like illness (General disorders) | 15 | 14
Tooth infection (Infections and infestations) | 10 | 16
Constipation (Gastrointestinal disorders) | 11 | 14
Urinary tract infection (Infections and infestations) | 14 | 10
Pruritus (Skin and subcutaneous tissue disorders) | 13 | 9
Sinusitis (Infections and infestations) | 7 | 14
Neck pain (Musculoskeletal and connective tissue disorders) | 12 | 8
Abdominal discomfort (Gastrointestinal disorders) | 14 | 4
Joint sprain (Injury, poisoning and procedural complications) | 7 | 11
Sciatica (Nervous system disorders) | 11 | 7
Fatigue (General disorders) | 12 | 5
Erythema (Skin and subcutaneous tissue disorders) | 15 | 1
Contusion (Injury, poisoning and procedural complications) | 5 | 10
Hypocalcaemia (Metabolism and nutrition disorders) | 5 | 10

LIMITATIONS AND CAVEATS:
The study showed an underexposure to calcitonin compared to what was expected from phase I trials.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days